CLINICAL TRIAL: NCT00642954
Title: A Phase I Study of Vorinostat in Combination With Lenalidomide and Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Vorinostat (MK-0683, SAHA [Suberoylanilide Hydroxamic Acid]) + Lenalidomide + Dexamethasone in Multiple Myeloma (MM) (MK-0683-074)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0683-074; 2007_511 (Other: Merck); 2007-001033-34 (EudraCT Number); MK-0683-074 (Other: Merck)
Record Dates: First submitted 2008-03-17; First posted 2008-03-25 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Vorinostat; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Level 1: Vorinostat 300 mg + lenalidomide 10 mg (Experimental): Participants will receive vorinostat 300 mg orally once-daily (QD) on Days 1-7 and Days 15-21; lenalidomide 10 mg orally QD on Days 1-21 and dexamethasone 40 mg orally QD on Days 1, 8, 15 and 22 of each 28-day cycle for up to 8 cycles. Qualified participants who don't have disease progression can continue treatment after 8 cycles at the same dose and schedule, until progressive disease or unacceptable toxicity.
  Interventions: Drug: Vorinostat; Drug: Lenalidomide; Drug: Dexamethasone
- Level 2: Vorinostat 400 mg + lenalidomide 10 mg (Experimental): Participants will receive vorinostat 400 mg orally QD on Days 1-7 and Days 15-21; lenalidomide 10 mg orally QD on Days 1-21 and dexamethasone 40 mg orally QD on Days 1, 8, 15 and 22 of each 28-day cycle for up to 8 cycles. Qualified participants who don't have disease progression can continue treatment after 8 cycles at the same dose and schedule, until progressive disease or unacceptable toxicity.
  Interventions: Drug: Vorinostat; Drug: Lenalidomide; Drug: Dexamethasone
- Level 3: Vorinostat 400 mg + lenalidomide 15 mg (Experimental): Participants will receive vorinostat 400 mg orally QD on Days 1-7 and Days 15-21; lenalidomide 15 mg orally QD on Days 1-21 and dexamethasone 40 mg orally QD on Days 1, 8, 15 and 22 of each 28-day cycle for up to 8 cycles. Qualified participants who don't have disease progression can continue treatment after 8 cycles at the same dose and schedule, until progressive disease or unacceptable toxicity.
  Interventions: Drug: Vorinostat; Drug: Lenalidomide; Drug: Dexamethasone
- Level 4: Vorinostat 400 mg + lenalidomide 20 mg (Experimental): Participants will receive vorinostat 400 mg orally QD on Days 1-7 and Days 15-21; lenalidomide 20 mg orally QD on Days 1-21 and dexamethasone 40 mg orally QD on Days 1, 8, 15 and 22 of each 28-day cycle for up to 8 cycles. Qualified participants who don't have disease progression can continue treatment after 8 cycles at the same dose and schedule, until progressive disease or unacceptable toxicity.
  Interventions: Drug: Vorinostat; Drug: Lenalidomide; Drug: Dexamethasone
- Level 5: Vorinostat 400 mg + lenalidomide 25 mg (Experimental): Participants will receive vorinostat 400 mg orally QD on Days 1-7 and Days 15-21; lenalidomide 25 mg orally QD on Days 1-21 and dexamethasone 40 mg orally QD on Days 1, 8, 15 and 22 of each 28-day cycle for up to 8 cycles. Qualified participants who don't have disease progression can continue treatment after 8 cycles at the same dose and schedule, until progressive disease or unacceptable toxicity.
  Interventions: Drug: Vorinostat; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Vorinostat — Vorinostat 300 mg or 400 mg QD via oral capsule on Days 1-7 and Days 15-21 of each 28-day cycle.
  Other Names: MK-0683; Suberoylanilide hydroxamic acid; Zolinza
Drug: Lenalidomide — Lenalidomide 10 mg, 15 mg, 20 mg or 25 mg QD via oral capsule on Days 1-21 of each 28-day cycle.
  Other Names: Revlimid
Drug: Dexamethasone — Dexamethasone 40 mg QD via oral tablet on Days 1, 8, 15 and 22 of each 28-day cycle.
  Other Names: Decadron

SUMMARY:
The purpose of this Phase I study of vorinostat in combination with lenalidomide and dexamethasone in participants with relapsed or refractory multiple myeloma is to determine the maximum tolerated dose (MTD) as estimated by the incidence of dose-limiting toxicities (DLTs) and recommended Phase 2 dose (RP2D) as estimated by the incidence of drug-related adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Is a male or female at least 18 years old
* Has relapsed or refractory MM and has had at least one prior therapy
* Female participants of childbearing potential must have 2 negative serum pregnancy tests prior to receiving the first dose of study drugs
* Female participants who can become pregnant must agree to use 2 separate forms of effective birth control at the same time, 4 weeks before, while taking, and for 4 weeks after stopping lenalidomide; post menopausal participants should be free from menses for >2 years, or are surgically sterilized
* Male participant agrees to use an adequate method of contraception for the duration of the study, even if the participant has undergone a successful vasectomy
* Male participants must agree to use a latex condom during sexual contact with a pregnant female or a female who can become pregnant; this is required for the duration of the study, and for 4 weeks after stopping therapy
* Has at least 3 weeks washout prior to treatment
* Is able to swallow capsules and is able to take or tolerate oral medications on a continuous basis

Exclusion Criteria:

* Has prior treatment with a histone deacetylase (HDAC) inhibitor
* Has prior allogenetic bone marrow transplant
* Has received intravenous antibiotics, antiviral, or antifungal agents within 2 weeks prior to the start of the study drug
* Uses illicit drugs, substance abuse or had a recent history (within the last year) of drug or alcohol abuse
* Is pregnant or breast feeding or expecting to have a baby during the course of the study
* Has human immunodeficiency virus (HIV) infection
* Has Hepatitis B/C infection
* Is currently receiving treatment for another type of cancer other than skin or cervical cancer that has not been in remission for 5 years or longer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-02-13 (Actual); Primary Completion 2012-09-03 (Actual); Study Completion 2013-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Siegel DS, Richardson P, Dimopoulos M, Moreau P, Mitsiades C, Weber D, Houp J, Gause C, Vuocolo S, Eid J, Graef T, Anderson KC. Vorinostat in combination with lenalidomide and dexamethasone in patients with relapsed or refractory multiple myeloma. Blood Cancer J. 2014 Feb 21;4(2):e182. doi: 10.1038/bcj.2014.1. PMID 24562384

RESULTS

PARTICIPANT FLOW:
Groups:
- Level 1: Vorinostat 300 mg + Lenalidomide 10 mg: Participants received vorinostat 300 mg orally once-daily (QD) on Days 1-7 and Days 15-21; lenalidomide 10 mg orally QD on Days 1-21 and dexamethasone 40 mg orally QD on Days 1, 8, 15 and 22 of each 28-day cycle for up to 8 cycles.
- Level 2: Vorinostat 400 mg + Lenalidomide 10 mg: Participants received vorinostat 400 mg orally QD on Days 1-7 and Days 15-21; lenalidomide 10 mg orally QD on Days 1-21 and dexamethasone 40 mg orally QD on Days 1, 8, 15 and 22 of each 28-day cycle for up to 8 cycles.
- Level 3: Vorinostat 400 mg + Lenalidomide 15 mg: Participants received vorinostat 400 mg orally QD on Days 1-7 and Days 15-21; lenalidomide 15 mg orally QD on Days 1-21 and dexamethasone 40 mg orally QD on Days 1, 8, 15 and 22 of each 28-day cycle for up to 8 cycles.
- Level 4: Vorinostat 400 mg + Lenalidomide 20 mg: Participants received vorinostat 400 mg orally QD on Days 1-7 and Days 15-21; lenalidomide 20 mg orally QD on Days 1-21 and dexamethasone 40 mg orally QD on Days 1, 8, 15 and 22 of each 28-day cycle for up to 8 cycles.
- Level 5: Vorinostat 400 mg + Lenalidomide 25 mg: Participants received vorinostat 400 mg orally QD on Days 1-7 and Days 15-21; lenalidomide 25 mg orally QD on Days 1-21 and dexamethasone 40 mg orally QD on Days 1, 8, 15 and 22 of each 28-day cycle. Treatment continued until progressive disease or unacceptable toxicity.
Period: Overall Study
Arm/Group | Level 1: Vorinostat 300 mg + Lenalidomide 10 mg | Level 2: Vorinostat 400 mg + Lenalidomide 10 mg | Level 3: Vorinostat 400 mg + Lenalidomide 15 mg | Level 4: Vorinostat 400 mg + Lenalidomide 20 mg | Level 5: Vorinostat 400 mg + Lenalidomide 25 mg
Started | 4 | 4 | 3 | 3 | 17
Completed | 0 | 0 | 0 | 0 | 1
Not Completed | 4 | 4 | 3 | 3 | 16
Not completed — Progressive Disease | 3 | 3 | 3 | 3 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Level 1: Vorinostat 300 mg + Lenalidomide 10 mg | Level 2: Vorinostat 400 mg + Lenalidomide 10 mg | Level 3: Vorinostat 400 mg + Lenalidomide 15 mg | Level 4: Vorinostat 400 mg + Lenalidomide 20 mg | Level 5: Vorinostat 400 mg + Lenalidomide 25 mg | Total
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 17 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.5 (4.7) | 58.5 (2.1) | 66.3 (6.1) | 55.7 (2.5) | 64.1 (7.2) | 63.5 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 1 | 7 | 13
  Male | 2 | 3 | 1 | 2 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose-Limiting Toxicities (DLTs)
Description: DLTs consisted of hematologic or non-hemtologic toxicities. Hematologic DLT was any grade (gr) 4 neutropenia lasting ≥7 days, gr 4 thrombocytopenia or gr 5 hematologic toxicity. Non-hematologic DLT was any gr 3, 4 or 5 non-hematologic toxicity with the exception of (1) gr 3 nausea, vomiting, diarrhea or dehydration not compliant with medical care, lasting <48 hours (2) gr 3 acidosis/alkalosis returning to ≤ gr 2 by 48 hours of medical care (3) gr 3 liver function test elevation without symptoms, lasting ≤5 days (4) Gr 3 amylase elevation without symptoms (5) Gr 3 hypocalcemia, hypokalemia, hypomagnesemia, hyponatremia or hyphosphatemia responding to medical care (6) Gr 3 hypercholeresterolemia or hypertriglyceridemia. A drug-related AE causing dose modification of study drug is also considered a DLT. Per protocol DLTs were analyzed in the first 28-day treatment cycle. The number of participants experiencing DLTs is reported here for all participants who got ≥1 dose of study drug.
Time Frame: Cycle 1 (Up to 28 days)
Population: All participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Level 1: Vorinostat 300 mg + Lenalidomide 10 mg | Level 2: Vorinostat 400 mg + Lenalidomide 10 mg | Level 3: Vorinostat 400 mg + Lenalidomide 15 mg | Level 4: Vorinostat 400 mg + Lenalidomide 20 mg | Level 5: Vorinostat 400 mg + Lenalidomide 25 mg
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 17
Participants | 0 | 0 | 0 | 0 | 1

2. Secondary Outcome: Number of Participants Experiencing Drug-Related Adverse Events (AEs)
Description: An AE was defined as any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product. Any worsening of a pre-existing condition which is temporally associated with the use of the Sponsor's product is also an AE. An AE was considered related to a drug as determined by the investigator based on exposure (evidence of exposure to drug), time course (time of AE onset versus drug-induced effect), likely cause (AE etiology related or un-related to drug), de-challenge (drug dose reduction/discontinuation) or re-challenge (drug re-exposure). Per protocol participants experiencing drug-related AEs were analyzed at the time of the protocol-specified final statistical analysis with a 3-September (Sep)-2012 data cut-off. The number of participants experiencing drug-related AEs is reported here for all participants who got ≥1 dose of study drug.
Time Frame: Up to ~55 months (through pre-specified final statistical analysis cut-off date of 3-Sep-2012)
Population: All participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Level 1: Vorinostat 300 mg + Lenalidomide 10 mg | Level 2: Vorinostat 400 mg + Lenalidomide 10 mg | Level 3: Vorinostat 400 mg + Lenalidomide 15 mg | Level 4: Vorinostat 400 mg + Lenalidomide 20 mg | Level 5: Vorinostat 400 mg + Lenalidomide 25 mg
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 17
Participants | 2 | 3 | 3 | 3 | 17

3. Other Pre Specified Outcome: Number of Participants Experiencing Best Overall Response Determined by Complete Response (CR), Near Complete Response (NCR), Very Good Partial Response (VGPR), Partial Response (PR), Minimal Response (MR), Stable Disease (SD) or Progressive Disease (PD)
Description: Best overall tumor response consisted of CR (negative M-protein immunofixation [IF], <5% bone marrow [BM] plasma cells, no soft tissue plasmacytomas [STP]), NCR (positive M-protein IF, <5% BM plasma cells, no STP), VGPR (≥90% M-protein decrease, <5% BM plasma cells, no STP), PR (≥50% M-protein, BM plasma cells, STP decrease), MR (25-49% M-protein, BM plasma cells, STP decrease), SD (<25% decrease-25% increase in M-protein, BM plasma cells; <25% decrease-increase in definite STP) or PD (≥25% M-protein, BM plasma cells increase; new STP, lesions). Per protocol participants experiencing best overall response by CR, NCR, VGPR, PR, MR, SD or PD were analyzed as a single prespecified analysis at the time of protocol-specified final statistical analysis with a 3-Sep-2012 data cut-off. The number of participants experiencing best overall response by CR, NCR, VGPR, PR, MR, SD or PD is reported here for all participants who got ≥1 dose of study drug and had a post baseline efficacy assessment.
Time Frame: Up to ~55 months (through pre-specified final statistical analysis cut-off date of 3-Sep-2012)
Population: All participants who received ≥1 dose of study treatment and had a post baseline efficacy assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Level 1: Vorinostat 300 mg + Lenalidomide 10 mg | Level 2: Vorinostat 400 mg + Lenalidomide 10 mg | Level 3: Vorinostat 400 mg + Lenalidomide 15 mg | Level 4: Vorinostat 400 mg + Lenalidomide 20 mg | Level 5: Vorinostat 400 mg + Lenalidomide 25 mg
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 16
Participants
  CR | 0 | 0 | 0 | 0 | 1
  NCR | 0 | 1 | 0 | 0 | 0
  VGPR | 1 | 0 | 0 | 1 | 2
  PR | 1 | 1 | 0 | 1 | 5
  MR | 0 | 0 | 1 | 0 | 2
  SD | 1 | 1 | 1 | 0 | 5
  PD | 1 | 1 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to ~66 months (through database cut-off date of 20-August-2013)
Description: Safety was analyzed in all participants who received ≥1 dose of study drug. Per protocol disease progression of cancer under study was not considered an AE unless considered related to study drug. Therefore Medical Dictionary for Regulatory Activities (MedDRA) preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | Level 1: Vorinostat 300 mg + Lenalidomide 10 mg | Level 2: Vorinostat 400 mg + Lenalidomide 10 mg | Level 3: Vorinostat 400 mg + Lenalidomide 15 mg | Level 4: Vorinostat 400 mg + Lenalidomide 20 mg | Level 5: Vorinostat 400 mg + Lenalidomide 25 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/4 | 0/3 | 0/3 | 3/17
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/4 | 1/3 | 2/3 | 8/17
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 3/3 | 3/3 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level 1: Vorinostat 300 mg + Lenalidomide 10 mg (N=4) | Level 2: Vorinostat 400 mg + Lenalidomide 10 mg (N=4) | Level 3: Vorinostat 400 mg + Lenalidomide 15 mg (N=3) | Level 4: Vorinostat 400 mg + Lenalidomide 20 mg (N=3) | Level 5: Vorinostat 400 mg + Lenalidomide 25 mg (N=17)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level 1: Vorinostat 300 mg + Lenalidomide 10 mg (N=4) | Level 2: Vorinostat 400 mg + Lenalidomide 10 mg (N=4) | Level 3: Vorinostat 400 mg + Lenalidomide 15 mg (N=3) | Level 4: Vorinostat 400 mg + Lenalidomide 20 mg (N=3) | Level 5: Vorinostat 400 mg + Lenalidomide 25 mg (N=17)
Anaemia (Blood and lymphatic system disorders) | 4 (11) | 1 (2) | 1 (8) | 3 (4) | 9 (28)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (10)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (9)
Neutropenia (Blood and lymphatic system disorders) | 2 (7) | 2 (3) | 1 (8) | 2 (11) | 6 (37)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (9) | 2 (4) | 1 (8) | 1 (1) | 12 (70)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breath odour (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (5) | 2 (2) | 1 (3) | 7 (20)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 6 (14)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-tussive vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (10)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 11 (60)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device complication (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 4 (6)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia primary atypical (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (4) | 1 (5) | 5 (7)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bone fragmentation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Electric shock (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 3 (9)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (4) | 1 (1) | 1 (1) | 2 (9)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (23)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood magnesium decreased (Investigations) | 3 (5) | 0 (0) | 1 (1) | 2 (2) | 2 (4)
Blood phosphorus decreased (Investigations) | 1 (5) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (9)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (5)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (8)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (4)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 4 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (23)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (9)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (6) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 1 (2) | 0 (0) | 3 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 5 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (2) | 2 (2) | 7 (13)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (11)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (1) | 1 (1) | 0 (0) | 4 (5)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (20)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (6)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (16)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Mood altered (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (3) | 1 (2) | 1 (1) | 7 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (15)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (7)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.